CLINICAL TRIAL: NCT02706535
Title: A Single Center, Two Part, Randomized, Open Label Cross-over Study to Evaluate the Effect of Itraconazole and Rifampicin on the Pharmacokinetics of GSK525762 in Healthy Female Subjects of Non Child Bearing Potential
Brief Title: A Cross-over Study to Evaluate the Effect of Itraconazole and Rifampicin on the Pharmacokinetics (PK) of GSK525762 in Healthy Female Subjects of Non Child Bearing Potential
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 204946
Record Dates: First submitted 2016-03-07; First posted 2016-03-11 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Drug Interactions; Neoplasms
Keywords: Itraconazole; Rifampicin; Pharmacokinetics; Cross-over
MeSH Terms: conditions — Neoplasms | interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 Cohort 1 (Experimental): Subjects will receive a single dose of GSK525762 10 mg on Day 1 followed by 200 mg Itraconazole two times a day (BID) on Day 3. On Day 4 to Day 6 inclusive subjects will receive a single dose of itraconazole 200 mg in the morning. On Day 7 subjects will receive a single dose of GSK525762 5 mg one hour after receiving 200 mg dose of itraconazole. On day 8 and 9 subjects will receive a single dose of 200 mg itraconazole in the morning.
  Interventions: Drug: GSK525762 Besylate Tablets; Drug: Itraconazole 200 mg
- Part 1 Cohort 2 (Experimental): Subjects will receive a single dose of GSK525762 10 mg on day 1 followed by 200 mg Itraconazole BID on day 3. On day 4 to day 6 inclusive subjects will receive a single dose of itraconazole 200 mg in the morning. On day 7 subjects will receive a single dose of GSK525762 5 mg or GSK525762 10 mg one hour after receiving 200 mg dose of itraconazole. On day 8 and 9 subjects will receive a single dose of 200 mg itraconazole in the morning.
  Interventions: Drug: GSK525762 Besylate Tablets; Drug: Itraconazole 200 mg
- Part 2 (Experimental): Subjects will receive a single dose of GSK525762 10 mg on day 1. From day 3 to 17 inclusive, subjects will receive a single dose of 600 mg rifampicin in fasting conditions. On day 18 subjects will receive single dose of GSK525762 either 20 or 30 mg along with 600 mg dose of rifampicin. On day 19 subjects will receive a single dose of rifampicin 600 mg.
  Interventions: Drug: GSK525762 Besylate Tablets; Drug: Rifampicin 300 mg

INTERVENTIONS:
Drug: GSK525762 Besylate Tablets — GSK525762 is available as a film-coated, white to slightly colored round, biconvex tablets with no markings. It is available in unit dose strength of 5 mg.
Drug: Itraconazole 200 mg — Itraconazole is available as a clear yellow solution with unit dose strength of 10 mg/mL
  Arms: Part 1 Cohort 1; Part 1 Cohort 2
Drug: Rifampicin 300 mg — Rifampicin is available as a red capsule with printed markings and as a 300 mg unit dose strength.
  Arms: Part 2

SUMMARY:
This is a Phase I, single center, two-part, randomized, open label, cross-over study. Part 1 of this study will evaluate the PK, safety, and tolerability of GSK525762 when administered alone and when co-administered following repeat dosing of itraconazole, a known strong inhibitor of Cytochrome P450 3A4 (CYP3A4) and a Para-glycoprotein (Pgp) inhibitor. Part 1 will consist of 2 Cohorts with preliminary PK and safety data obtained from Cohort 1 informing Cohort 2. Part 2 (one Cohort) of the study will evaluate the PK, safety, and tolerability of GSK525762 when administered alone and when co-administered following repeat dosing of rifampicin, a known potent inducer of CYP3A4. In vitro inhibition data indicate CYP3A4 may be the major route of clearance for GSK525762 and co-administration of drug therapies which modulate CYP3A4 (i.e.CYP3A4 inhibitors and inducers) is likely to alter the exposure of GSK525762 (i.e. increase or decrease exposure, respectively). The data generated from this current study to justify exclusion criteria on concomitant medications which affect CYP3A4 or Pgp and also inform potential dose modification in case of co-administration with medication affecting CYP3A4 activity. All subjects will undergo a screening visit within 28 days of the first dose of study drug followed by one treatment period and a follow-up visit 7-10 days after the last dose of GSK525762. Subjects in Part 1 will participate in the study for up to 45 days and subjects in Part 2 will participate for up to 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, and laboratory tests.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body Weight >=45 Kilograms (Kg) and body mass index within the range 18.0 - 29.9 Kilograms/squared meter (kg/m^2) (inclusive) at time of screening.
* Only female subjects of non child bearing potential are eligible for screening; men are not eligible for this study. Female subjects: are eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test at screening and serum or urine hCG prior to dosing), is not lactating, and lacks reproductive potential, defined as:

  * Pre-menopausal females with one of the following:

    1. Documented tubal ligation
    2. Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion
    3. Hysterectomy
    4. Documented Bilateral Oophorectomy
  * Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)].
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* ALT and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Cardiac abnormalities as evidenced by any of the following:

  * History or current untreated clinically significant uncontrolled arrhythmias.
  * Clinically significant conduction abnormalities or arrhythmias, subjects with Bundle Branch Block
  * Presence of cardiac pacemaker
  * History or evidence of current >=Class II congestive heart failure as defined by New York Heart Association (NYHA).
  * History of acute coronary syndromes (including unstable angina and myocardial infarction), coronary angioplasty, or stenting.
* Any of the following ECG findings:

Baseline QT duration corrected for heart rate by Fridericia's formula (QTcF) interval >450 miliseconds.

* History of major gastrointestinal bleeding within the last 6 months. Any evidence of active gastrointestinal bleeding excludes the subject.
* An unwillingness to abstain from all concomitant medications (excluding acetaminophen).
* History of regular alcohol consumption within 3 months of the study defined as:

  •An average weekly intake of >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 millilitre [ml]) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* A positive test for alcohol at screening or on admission to the clinical unit.
* A positive urine drug test at screening or on admission to the clinical unit.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* An unwillingness to abstain from caffeine- and xantheine- containing products for 24 hours prior to GSK525762 dosing until collection of the final PK sample during each PK session.
* An unwillingness to abstain from ingestion of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos within 7 days prior to the first dose of study treatment(s) or until the end of the study.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longest).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-06 (Actual)

PRIMARY OUTCOMES:
Part 1: Area under the plasma concentration-time curve (AUC) from pre dose to time 't' (AUC[0-t]) and pre dose to infinite time (AUC[0-infinity]) of GSK525762 and metabolites in the presence and absence of itraconazole | Day 1: Pre dose, 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 8 hr, 12 hr, 24 hr , 36 hr, and 48 hr post dose. Day 7:Pre dose, 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 8 hr, 12 hr, 24 hr, 36 hr, 48 hr and 72 hr.
Part 1: Maximum plasma concentration (Cmax) of GSK525762 and metabolites in the presence and absence of itraconazole | Day1 (Pre dose and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 8 hr, 12 hr, 24 hr, 36 hr, and 48 hr post dose) and Day7 (Pre dose and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 8 hr, 12 hr, 24 hr, 36 hr, 48 hr and 72 hr post dose) of each cohort
Part 1: Time to maximum plasma concentration (tmax) of GSK525762 and metabolites in the presence and absence of itraconazole | Day1 (Pre dose, 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 8 hr, 12 hr, 24 hr , 36 hr, and 48 hr) and Day7 (Pre dose, 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 8 hr, 12 hr, 24 hr, 36 hr, 48 hr and 72 hr) of each cohort
Part 2: (AUC[0-t]) and (AUC[0-infinity]) of GSK525762 and metabolites in the presence and absence of rifampicin | Blood samples will be collected on Day1 and Day 18 at Pre dose, 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 8 hr, 12 hr, 24 hr (Day 19), 36 hr, and 48 hr (Day 20) post dose
Part 2: Cmax of GSK525762 and metabolites in the presence and absence of rifampicin | Blood samples will be collected on Day 1 and Day 18 at Pre dose, 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 8 hr, 12 hr, 24 hr (Day 19), 36 hr, and 48 hr (Day 20) post dose
Part 2: tmax of GSK525762 and metabolites in the presence and absence of rifampicin | Blood samples will be collected on Day 1 and Day 18 at Pre dose, 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 8 hr, 12 hr, 24 hr (Day 19), 36 hr, and 48 hr (Day 20) post dose

SECONDARY OUTCOMES:
Part 1: Number of subjects with adverse event (AE) and serious adverse event (SAE) | Up to 45 days
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement will be categorized as SAE
Part 1: Number of subjects having abnormal haematology parameters as a measure of safety. | Up to 45 days
  Blood samples will be collected at screening, pre dose (Day 1), and post dose on Day 3,Day 6 and at follow-up visit to analyze platelet counts, red blood cells (RBC) count, white blood cells (WBC) count (absolute), haemoglobin, hematocrit and differential WBC count ( neutrophils, lymphocytes, monocytes, eosinophils, and basophils).
Part 1: Number of subjects having abnormal clinical chemistry parameters as a measure of safety | Up to 45 days
  Blood samples will be collected at screening, pre dose (Day 1), and post dose on Day 3,Day 6 and at follow-up visit to analyze blood urea nitrogen (BUN), creatinine, glucose (fasting), sodium, c peptide, potassium, chloride, magnesium, ionized calcium, aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT), alkaline phosphatase (ALP) levels, gamma-glutamyltransferase (GGT), total and direct bilirubin, total carbon dioxide, total protein and albumin
Part 1: Number of subjects having abnormal urine parameters (using dipstick test) as a measure of safety | Up to 45 days
  Urine samples will be collected at screening, pre dose (Day 1), and post dose on Day 3,Day 6 and at follow-up visit to analyze specific gravity, pH, glucose, protein, blood and ketone bodies by dipstick method, microscopic examination (if blood or protein is abnormal) WBCs, RBCs, hyaline casts, granular casts and cellular casts.
Part 1: Electrocardiogram (ECG) assessment as a measure of safety and tolerability | Up to 45 days
  ECGs will be measured in supine position after 5 minutes rest using a standard 12-lead ECG machine that automatically calculates the HR and measures PR, QRS, QT and QTcF intervals.
Part 1: Blood pressure assessment as a safety measure. | Up to 45 days
  Systolic and diastolic blood pressure will be measured on each day in supine or semi-supine position after 5 minutes rest.
Part 1: Heart rate assessment as a safety measure. | Up to 45 days
  Heart rate will be measured on each day in supine or semi-supine position after 5 minutes rest.
Part 2: Number of subjects with adverse event (AE) and serious adverse event (SAE) | Up to 56 days
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement will be categorized as SAE.
Part 2: Number of subjects having abnormal haematology parameters as a measure of safety. | Up to 56 days
  Blood samples will be collected at screening, pre dose (Day 1), and post dose on Day 3,Day 4, Day 17 and at follow-up to analyze platelet counts, RBC count, WBC count (absolute), haemoglobin, hematocrit and differential WBC count ( neutrophils, lymphocytes, monocytes, eosinophils, and basophils).
Part 2: Number of subjects having abnormal clinical chemistry parameters as a measure of safety. | Up to 56 days
  Blood samples will be collected at screening, pre dose (Day 1), and post dose on Day 3,Day 4, Day 17 and at follow-up visit to analyze BUN, creatinine, glucose (fasting), sodium, c peptide, potassium, chloride, magnesium, ionized calcium, AST/SGOT, ALT/SGPT, ALP levels, GGT, total and direct bilirubin, total carbon dioxide, total protein and albumin
Part 2: Number of subjects having abnormal urine parameters (using dipstick test) as a measure of safety. | Up to 56 days
  Urine samples will be collected at screening, pre dose (Day 1), and post dose on Day 3,Day 4, Day 17 and at follow-up visit to analyze specific gravity, pH, glucose, protein, blood and ketone bodies by dipstick method, microscopic examination (if blood or protein is abnormal) WBCs, RBCs, hyaline casts, granular casts and cellular casts.
Part 2: ECG assessment as a measure of safety and tolerability. | Up to 56 days
  On Day 1 and Day 18 ECGs will be measured in supine position after 5 minutes rest at screening, pre-dose, 1 hr, 24 hr and 48 hrs.
Part 2: Blood pressure assessment as a safety measure. | Up to 56 days
  Systolic and diastolic blood pressure will be measured on each day in supine or semi-supine position after 5 minutes rest.
Part 2: Heart rate assessment as a safety measure. | Up to 56 days
  Heart rate will be measured on each day in supine or semi-supine position after 5 minutes rest.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20724

REFERENCES:
- [Background] Riddell K, Patel A, Collins G, Zhou Y, Schramek D, Kremer BE, Ferron-Brady G. An Adaptive Physiologically Based Pharmacokinetic-Driven Design to Investigate the Effect of Itraconazole and Rifampicin on the Pharmacokinetics of Molibresib (GSK525762) in Healthy Female Volunteers. J Clin Pharmacol. 2021 Jan;61(1):125-137. doi: 10.1002/jcph.1711. Epub 2020 Aug 20. PMID 32820548